CLINICAL TRIAL: NCT07316790
Title: Comparative Evaluation Study of Retro Discal Tissue Injection Arthroscopically Versus Ultrasound Guide Injection
Brief Title: Evaluation Study of Retro Discal Tissue Injection Arthroscopically Versus Ultrasound Guide Injection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wajmah Sayed Karim Al Sayed, Principal Investigator, PhD Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: arthroscope versus ultrasound
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Arthroscope

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic Retrodiscal Tissue Injection (Experimental): Arthroscopic Retrodiscal Tissue Injection
  Interventions: Procedure: Arthroscopic retrodiscal tissue injection
- Ultrasound-Guided Retrodiscal Tissue Injection (Active Comparator): Ultrasound-Guided Retrodiscal Tissue Injection
  Interventions: Procedure: Ultrasound-guided retrodiscal tissue injection

INTERVENTIONS:
Procedure: Arthroscopic retrodiscal tissue injection — Arthroscopic retrodiscal tissue injection
  Arms: Arthroscopic Retrodiscal Tissue Injection
Procedure: Ultrasound-guided retrodiscal tissue injection — Ultrasound-guided retrodiscal tissue injection
  Arms: Ultrasound-Guided Retrodiscal Tissue Injection

SUMMARY:
A comparative evaluation study of arthroscopic retrodiscal tissue injection versus ultrasound-guided injection in temporomandibular joint disorders aims to assess differences in pain relief, functional improvement, and clinical outcomes between an invasive and a minimally invasive delivery technique. Arthroscopic injection allows direct visualization of intra-articular structures, accurate targeting of the retrodiscal tissues, and simultaneous management of associated pathology such as synovitis or adhesions, which may enhance therapeutic outcomes in advanced internal derangement. In contrast, ultrasound-guided injection offers a less invasive, cost-effective, and outpatient-based approach with improved accuracy over blind techniques, making it suitable for early or moderate cases. While both methods are effective in reducing pain and improving mouth opening and jaw function, arthroscopic injection may provide superior results in patients requiring diagnostic confirmation and mechanical intervention, whereas ultrasound-guided injection offers comparable symptomatic improvement with lower procedural morbidity and resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years with symptomatic TMJ disorder/internal derangement (unilateral or bilateral)
* TMJ pain at rest and/or during function for ≥ 3 months
* Clinical diagnosis consistent with disc displacement with or without reduction (with or without MRI confirmation, if included in the protocol)
* Baseline pain intensity ≥ 4/10 on VAS or NRS
* Limitation of mouth opening or functional impairment (e.g., maximum mouth opening ≤ 35 mm or pain-related limitation)
* Failed or insufficient response to conservative therapy for ≥ 4-6 weeks (e.g., soft diet, NSAIDs, splint therapy, physiotherapy)
* Ability to provide informed consent and comply with scheduled follow-up visits

Exclusion Criteria:

* Previous TMJ surgery (arthroscopy or arthrotomy) on the study side or TMJ injection within the last 3-6 months
* TMJ ankylosis, fracture, tumor, or active infection
* Primary inflammatory arthropathy (e.g., rheumatoid arthritis, gout, psoriatic arthritis) or systemic connective tissue disease affecting the TMJ
* Significant degenerative joint disease (advanced osteoarthritis) if the study focuses on internal derangement or soft tissue pathology
* Severe skeletal or dentofacial deformity requiring orthognathic surgery during the study period
* Pregnancy or lactation
* Bleeding disorders, platelet disorders, or anticoagulant therapy that cannot be safely managed (particularly relevant for PRP injections)
* Known allergy or contraindication to the planned injectate or local anesthetic
* Severe uncontrolled systemic disease (ASA III-IV) or inability to tolerate anesthesia or sedation (for arthroscopy arm)
* Active psychiatric or neurologic condition that may impair accurate pain reporting or follow-up compliance

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-13 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (VAS) | Baseline → 2 months (early outcome) Baseline → 6 months (mid-term outcome)
  Change in TMJ pain score measured on a 10-cm Visual Analogue Scale (0 = no pain, 10 = worst pain) from baseline to 3 months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Niveen AL Asker, Prof, Principal Investigator — Cairo University; Niveen AL Asker, Prof, Study Director — Cairo University
Locations (1):
- facility of Dentistry, Cairo, Old Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) generated during this study will be made available to other researchers upon reasonable request. The shared IPD will include baseline demographic data, clinical diagnosis, intervention allocation, pain scores (VAS), maximum mouth opening measurements, and follow-up outcome data at predefined time points. All shared data will be anonymized to ensure participant confidentiality, and no direct identifiers will be disclosed. Data will be available after publication of the primary study results and may be used for academic and non-commercial research purposes following approval by the study investigators.
Supporting Information: Study Protocol, ICF
Time Frame: by the end of May 2026 will be available
Access Criteria: throw the free publication

REFERENCES:
- [Result] Cha YH, O J, Park JK, Yang HM, Kim SH. Ultrasound-guided versus blind temporomandibular joint injections: a pilot cadaveric evaluation. Int J Oral Maxillofac Surg. 2019 Apr;48(4):540-545. doi: 10.1016/j.ijom.2018.09.002. Epub 2018 Oct 2. PMID 30287106
- [Result] Lopez JP, Orjuela MP, Gonzalez LV, Peraza-Labrador AJ, Diaz-Baez D. Comparison of the Clinical Effectiveness of Intra-Articular Injection with Different Substances After TMJ Arthroscopy: A Systematic Review and Meta-Analysis. J Maxillofac Oral Surg. 2024 Apr;23(2):261-270. doi: 10.1007/s12663-023-02047-7. Epub 2023 Dec 12. PMID 38601255